CLINICAL TRIAL: NCT03628014
Title: A Measure of the Effects of the Hospital Elder Life Program at the Jewish General Hospital: a Pre-post Intervention Study
Brief Title: The Hospital Elder Life Program at the Jewish General Hospital
Acronym: HELP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties and bad data quality
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal Investigator, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CODIM-MBM-17-182
Record Dates: First submitted 2018-02-01; First posted 2018-08-14 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Delirium; Fall Injury; Mortality
Keywords: older, hospital, program
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Other): The HELP Program is a comprehensive inpatient-care program that ensures optimal care for older adults in the hospital by using trained volunteers that do specific activities to help prevent or maintain functional decline.
  Interventions: Other: Inpatient-care program

INTERVENTIONS:
Other: Inpatient-care program — Patients enrolled in the Hospital Elder Life Program can receive four types of personalized volunteer-led interventions based on the needs identified by the care team. These interventions include:
  * Daily orientation and visiting program
  * Basic active movements
  * Meal assistance
  * Recreational activities

SUMMARY:
Older patients (i.e.; ≥ 65 years) with a hip fracture, and who are admitted to orthopedics for surgery are particularly at risk of adverse health events such as delirium, recurrent falls and prolonged hospital stay caused by their frailty status. The Hospital Elder Life Program (HELP) is a comprehensive inpatient-care program that ensures optimal care for older adults in the hospital and, thus, might reduce the incidence of postoperative adverse health events. The overall objective of this study is to examine in a quantitative fashion the effects of the HELP program on adverse health events in geriatric inpatients admitted to the orthopedic ward at JGH for surgery after a hip fracture.

DETAILED DESCRIPTION:
Delirium and mobility impairment with high risk of falls are important medical complications after a hip surgery. More than 95% of hip fractures are caused by falling and the risk of a new fall after a hip surgery may be up to 50%. Both postoperative delirium and fall are associated with increased length of stay and high perioperative mortality.

The Hospital Elder Life Program (HELP) is a comprehensive inpatient-care program that ensures optimal care for older adults in the hospital. The primary goals of the HELP program are:

Maintaining cognitive and physical functioning of high risk older adults throughout hospitalization, maximizing independence at discharge, assisting with the transition from hospital to home, and preventing unplanned hospital readmissions. These goals have been accomplished using a multicomponent intervention strategy. In addition to targeted interdisciplinary geriatric assessment, the program uses an innovative volunteer model to provide personal, supportive attention to vulnerable older inpatients.

ELIGIBILITY:
Inclusion Criteria:

* age 65 and over
* admitted to orthopedic ward for hip surgery after a fracture

Exclusion Criteria:

* younger than 65 years of age
* palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Presence of delirium after a hip surgery | 24 hours after surgery
  As measure will be used the CAM ( Confusion Assessment Method)

SECONDARY OUTCOMES:
Number of falls before having a hip fracture | Up to one month
  The number of falls are recorded in medical chart
In-hospital mortality | Up to one month
  Mortality during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada